CLINICAL TRIAL: NCT03834935
Title: Efficacy of Topical Pimecrolimus in the Treatment of Pityriasis Alba: A Randomized Placebo-controlled Trial
Brief Title: Efficacy of Topical Pimecrolimus in the Treatment of Pityriasis Alba
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: St Joseph University, Beirut, Lebanon (Other)
Responsible Party: Principal Investigator, elio kechichian, Principal investigator, MD, St Joseph University, Beirut, Lebanon
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: USJDERM1
Record Dates: First submitted 2019-02-06; First posted 2019-02-08 (Actual); Last update posted 2019-02-11 (Actual); Status verified 2019-02

CONDITIONS: Pityriasis Alba
Keywords: pityriasis alba; treatment; topical calcineurin inhibitor
MeSH Terms: conditions — Dandruff | interventions — pimecrolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: investigators and patients will be blinded to treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pim (Experimental): 20 patients receiving topical Elidel (pimecrolimus 1%) bid on the affected area for 9 weeks.Sunscreens will not be indicated, and hygienic habits will not be changed.
  Interventions: Drug: Elidel (pimecrolimus 1%)
- Pl (Placebo Comparator): 20 patients receiving placebo (control group), cold cream bid on the affected area for 9 weeks.Sunscreens will not be indicated, and hygienic habits will not be changed.
  Interventions: Drug: Cold Cream

INTERVENTIONS:
Drug: Elidel (pimecrolimus 1%) — topical application of product on all lesions, twice daily. Sunscreen will not be indicated, and hygienic habits will not be changed
  Arms: Pim
Drug: Cold Cream — Topical application on all lesions, twice daily. Sunscreen will not be indicated, and hygienic habits will not be changed
  Arms: Pl

SUMMARY:
Pityriasis alba (PA) is a common benign skin disorder, that usually affects children and adolescents of darker phototypes. A history of atopic dermatitis is a well-known risk factor, and PA may be a minor manifestation of atopic dermatitis, although it can occur in nonatopic individuals as well. The objective is to evaluate the effect of topical pimecrolimus in the treatment of treatment of PA

DETAILED DESCRIPTION:
Background and Rationale:

Pityriasis alba (PA) is a common benign skin disorder, that usually affects children and adolescents of darker phototypes. PA usually manifests as erythematous lesions followed by smooth scales with residual characteristic pruritic or non-pruritic ill-defined hypopigmented patches, that typically occur on the upper part of the body, especially the face. A history of atopic dermatitis is a well-known risk factor, and PA may be a minor manifestation of atopic dermatitis, although it can occur in nonatopic individuals as well. It is thought to represent nonspecific dermatitis with residual post-inflammatory hypopigmentation. Sun exposure is a triggering and accentuating factor.

PA is a common reason for dermatologic consultation due to its chronic course, frequent relapses and cosmetic appearance. Spontaneous healing occurs in several months to few years, therefore impacting the quality of life. Emollients and mild-potency topical steroids are the mainstay of treatment, with a potential risk of skin atrophy and hypopigmentation.

Pimecrolimus is a topical calcineurin inhibitor that prevents T-cell activation, approved for the treatment of atopic dermatitis, and proved efficacious for seborrheic dermatitis, without having the potential adverse effects of topical corticosteroids. Tacrolimus 0.1% ointment, another calcineurin inhibitor is an effective and safe treatment for PA, a similar efficacy of calcitriol and tacrolimus was shown after 9 weeks of treatment. An exploratory study evaluated the efficacy of pimecrolimus cream in the treatment of PA. To the best of our knowledge there is no randomized placebo-controlled trial in the literature proving the efficacy of pimecrolimus in PA.

Objective: To evaluate the effect of topical pimecrolimus in the treatment of treatment of PA

Hypothesis: Pimecrolimus is an efficacious, well-tolerated and safe treatment for pityriasis alba.

Trial design: A randomized placebo-controlled double blinded trial establishing the superiority of topical pimecrolimus 1% over placebo.

ELIGIBILITY:
Inclusion Criteria:

* Pityriasis alba Patients confirmed by a board certified dermatologist
* Age over 2 years
* Written informed consent signed by the patients or the legal guardians of patients younger than 18 years in the native language (Arabic)

Exclusion Criteria:

* Other concomitant dermatosis (except atopic dermatitis)
* Use of topical steroids, or topical agents other than emollients and sunscreen, in the last 4 weeks
* Known allergy to pimecrolimus
* Pregnant and nursing women

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-03-01 (Estimated); Primary Completion 2021-02-01 (Estimated); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of repigmentation of index lesions | 9 weeks
  Objective percentage of repigmentation the index lesion (the largest lesion) by image analysis software (ImageJ software will be used to measure the lesion reduction area after treatments)

SECONDARY OUTCOMES:
Pruritus and scaling | 3,6 and 9 weeks
  IGA 4 point-scale (0: none - 3: severe)
Investigator's repigmentation change | 3,6 and 9 weeks
  Clinical change is assessed by means of digital photographic registration (frontal, right, and left views). An independent observer clinically graded the global improvement as poor (0-25%), mild (26-50%), good (51-75%), and excellent (>75%).
patient satisfaction | 9 weeks
  (0: not satisfied, 1: satisfied, 2: very satisfied).
Adverse events | 3,6 and 9 weeks
  adverse events reporting

CONTACTS AND LOCATIONS:
Overall Officials: Josiane Helou, MD, Study Chair — Saint-Joseph University
Locations (1):
- Saint Joseph University, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: Undecided